CLINICAL TRIAL: NCT04844853
Title: High Resolution Electroencephalography Exploration of Tactile Prediction Development
Brief Title: Neural Correlates of Tactile Prediction
Acronym: DECODE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2020-A03208-31
Record Dates: First submitted 2021-04-02; First posted 2021-04-14 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-07

CONDITIONS: Neurodevelopmental Disorders; Premature Birth
MeSH Terms: conditions — Neurodevelopmental Disorders; Premature Birth | interventions — Electroencephalography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Preterm 2 (Experimental): 2-year-olds born prematurely
  Interventions: Device: electroencephalography; Device: Tactile stimulation
- Term 2 (Experimental): 2-year-olds born at term
  Interventions: Device: electroencephalography; Device: Tactile stimulation
- Typical 6 (Experimental): 6-year-olds with typical developement
  Interventions: Device: electroencephalography; Device: Tactile stimulation; Behavioral: Attention Network task (computerized); Behavioral: Head-toes-knees-schoulders; Behavioral: Laby 5-12; Behavioral: M-ABC 2; Behavioral: Stroop animals
- NDD 6 (Experimental): 6-year-olds with neurodevelopmental disorders
  Interventions: Device: electroencephalography; Device: Tactile stimulation; Behavioral: Attention Network task (computerized); Behavioral: Head-toes-knees-schoulders; Behavioral: Laby 5-12; Behavioral: M-ABC 2; Behavioral: Stroop animals

INTERVENTIONS:
Device: electroencephalography — 128-channel electroencephalography
  Other Names: EEG
Device: Tactile stimulation — Vibrotactile sequence on the forearm
Behavioral: Attention Network task (computerized) — Computer-based game challenging orienting and executive attention. The subject must chose which side an animal is going, using left and right buttons, depending on the validity of a cue and the congruency of flankers.
  Other Names: Child ANT, flankers task
  Arms: NDD 6; Typical 6
Behavioral: Head-toes-knees-schoulders — Following motor commands such as touch your head when they are congruent or incongruent.
  Other Names: HTKS
  Arms: NDD 6; Typical 6
Behavioral: Laby 5-12 — Test of motor planning using labyrinths
  Arms: NDD 6; Typical 6
Behavioral: M-ABC 2 — Test of motor functions using various subtests of gross and fine motor function.
  Arms: NDD 6; Typical 6
Behavioral: Stroop animals — Stroop test for preK children using animals instead of words
  Arms: NDD 6; Typical 6

SUMMARY:
This project aims to measure repetition suppression and tactile prediction using high-resolution electroencephalography in preschoolers, in order to describe the responses as a function of age, gestational age of birth and the presence of a neurodevelopmental disorder. We will include 100 children aged 2 or 6 years: 25 2-year-olds born prematurely, 25 2-year-olds born at term, 25 6-year-olds with typical development and 25 6-year-olds with neurodevelopmental disorders. We will perform several behavioral evaluations to analyze the results in view of the quality of development.

DETAILED DESCRIPTION:
We will include 100 children aged 2 or 6 years: 25 2-year-olds born prematurely, 25 2-year-olds born at term, 25 6-year-olds with typical development and 25 6-year-olds with neurodevelopmental disorders. Children will be recruited from local schools and institutions. Birth will be considered premature if children were born before 36 weeks of gestational age. Children will be considered as having neurodevelopmental disorder if they receive medical and/or paramedical care at the time of measurement for neurodevelopmental disorder, including autism spectrum disorder, attention deficit with or without hyperactivity, tics, learning disorders, but all participants must be attending school at the time of measurement.

Children will come to the lab for a 2 hours session with their parents, during which they will undergo movement, attention and executive functions evaluations. Parents will fill out questionnaires evaluating their child's executive functioning and sensory profile in home/everyday settings. Children will then be equipped with 128-channels electroencephalography and proposed two tests : a modified attention network task and a tactile prediction task.

We will calculate correlations between evoked potential amplitudes during the tactile prediction trials and inhibitory conflict trials. Results will be analysed in the light of age, gestational age at birth, ecological and psychometric evaluations, and neurodevelopmental status.

ELIGIBILITY:
Inclusion Criteria:

* Age 24 to 35 or 72 to 83 months
* Born prematurely or term, with or without neurodevelopmental disorders (see arms)
* Parental informed consent
* Attending school

Exclusion Criteria:

* Severe IQ deficit or language impairment
* Psychotropic medication

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-04-30 (Estimated); Study Completion 2023-09-30 (Estimated)

PRIMARY OUTCOMES:
Repetition suppression at 2 | 2 years
  Difference of tactile evoked potential amplitude between end and beginning of stimulation sequence
Repetition suppression at 6 | 6 years
  Difference of tactile evoked potential amplitude between end and beginning of stimulation sequence
Tactile prediction at 2 | 2 years
  Difference of amplitude between baseline and omission segment
Tactile prediction at 6 | 6 years
  Difference of amplitude between baseline and omission segment

CONTACTS AND LOCATIONS:
Locations (1):
- Comete U1075 Inserm Unicaen, Caen, France

IPD SHARING:
Plan to Share IPD: No